CLINICAL TRIAL: NCT01913665
Title: The Effect of Bifidobacterium Lactis and Inulin on Functional Constipation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Makbule Eren, Associate professor, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: not defined yet
Record Dates: First submitted 2013-07-30; First posted 2013-08-01 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Functional Constipation
MeSH Terms: interventions — Inulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- B.Lactis (Active Comparator): children with functional constipation
  Interventions: Other: B.lactis
- Inulin (Active Comparator): children with functional constipation
  Interventions: Other: Inulin
- B.Lactis+ınulin (Active Comparator): children with functional constipation
  Interventions: Other: B.Lactis +Inulin
- plasebo (Placebo Comparator): children with functional constipation
  Interventions: Other: Placebo

INTERVENTIONS:
Other: B.lactis
  Arms: B.Lactis
Other: Inulin
  Arms: Inulin
Other: B.Lactis +Inulin
  Arms: B.Lactis+ınulin
Other: Placebo
  Arms: plasebo

SUMMARY:
The aim of this study is to asses the effect of Bifidobacterium lactis and Inulin on functional constipation in children

ELIGIBILITY:
Inclusion Criteria:

* children with functional constipation over 3 years age
* below 18 years of age

Exclusion Criteria:

* Chronic gastrointestinal disease,
* hirschsprung disease,
* celiac disease,
* hypothyroids,
* neurological deficit,
* constipation treatment receiving children will be excluded

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
to compare defecation frequency between baseline and 4 th week of treatment | baseline and 4th week of intervention